CLINICAL TRIAL: NCT03456063
Title: A Phase III, Double-Blinded, Multicenter, Randomized Study Evaluating the Efficacy and Safety of Neoadjuvant Treatment With Atezolizumab or Placebo in Combination With Platinum-Based Chemotherapy in Patients With Resectable Stage II, IIIA, or Select IIIB Non-Small Cell Lung Cancer
Brief Title: A Study of Neoadjuvant Atezolizumab Plus Chemotherapy Versus Placebo Plus Chemotherapy in Patients With Resectable Stage II, IIIA, or Select IIIB Non-Small Cell Lung Cancer (IMpower030)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO40241; 2023-504209-35-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2018-03-05; First posted 2018-03-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Small-Cell Lung
MeSH Terms: interventions — atezolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed; Carboplatin; Cisplatin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Atezolizumab + platinum-based chemotherapy (Experimental): Neoadjuvant treatment will consist of 4 cycles; atezolizumab + platinum-based chemotherapy
  Platinum-based chemotherapy may include:
  * carboplatin + pemetrexed
  * carboplatin + nab-paclitaxel
  * cisplatin + pemetrexed
  * cisplatin + gemcitabine
  Post-operative adjuvant treatment will consist of 16-cycles of atezolizumab
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Nab-paclitaxel; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine
- Arm B: Placebo + platinum-based chemotherapy (Placebo Comparator): Neoadjuvant treatment will consist of 4 cycles; placebo + platinum-based chemotherapy
  Platinum-based chemotherapy may include:
  * carboplatin + pemetrexed
  * carboplatin + nab-paclitaxel
  * cisplatin + pemetrexed
  * cisplatin + gemcitabine
  Participants will receive best supportive care and monitoring after surgery
  Interventions: Drug: Placebo Comparator; Drug: Nab-paclitaxel; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab will be administered as intravenous (IV) infusion at a dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle (every 3 weeks) for 4 cycles during the neoadjuvant treatment phase
  Atezolizumab will be administered as IV infusion at a dose of 1200 milligrams (mg) every 3 weeks for 16 cycles during the post-operative adjuvant phase
  Other Names: Tecentriq
  Arms: Arm A: Atezolizumab + platinum-based chemotherapy
Drug: Placebo Comparator — Placebo will be administered as IV infusion at a dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle for 4 cycles during the neoadjuvant treatment phase
  Arms: Arm B: Placebo + platinum-based chemotherapy
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/m^2 will be administered intravenously on Days 1, 8, and 15 of each 21 day cycle for 4 cycles during the neoadjuvant treatment phase
  Other Names: Abraxane
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle for 4 cycles during the neoadjuvant treatment phase
  Other Names: Alimta
Drug: Carboplatin — Carboplatin initial target AUC of 6 mg/mL/min will be administered intravenously on Day 1 of each 21-day cycle for 4 cycles during the neoadjuvant treatment phase
Drug: Cisplatin — Cisplatin 75 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle for 4 cycles during the neoadjuvant treatment phase
Drug: Gemcitabine — Gemcitabine 1250 mg/m^2 will be administered intravenously on Day 1 and 8 of each 21-day cycle for 4 cycles during the neoadjuvant treatment phase
  Other Names: Gemzar

SUMMARY:
This is a randomized, double-blinded study designed to evaluate the efficacy, safety, pharmacokinetics, and immunogenicity of neoadjuvant treatment with atezolizumab (MPDL3280A) or placebo in combination with platinum-based chemotherapy in participants with resectable Stage II, IIIA, or select IIIB non-small cell lung cancer (NSCLC) followed by open-label adjuvant/postoperative atezolizumab or best supportive care and monitoring.

ELIGIBILITY:
Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Histologically or cytologically confirmed, resectable Stage II, IIIA, or Select IIIB (T3N2 only) NSCLC of squamous or non-squamous histology. Staging should be based on the 8th edition of the AJCC/UICC staging system
* Evaluation by an attending thoracic surgeon to confirm eligibility for an R0 resection with curative intent
* Adequate pulmonary and cardiac function to undergo surgical resection
* Measurable disease as defined by RECIST v1.1
* Adequate hematologic and end organ function
* Negative HIV test at screening
* Negative for active HBV and HCV at screening
* Adequate tissue for PD-L1 IHC assessment

Exclusion criteria:

* NSCLC with histology of large cell neuroendocrine carcinoma or sarcomatoid carcinoma
* Mixed NSCLC and small cell lung cancer histology
* Any prior therapy for lung cancer
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated expected curative outcome
* Non-squamous NSCLC histology with activating ALK and EGFR mutation
* Pregnant or lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or evidence of active of active pneumonitis on screening chest Computed Tomography (CT) scan
* Prior treatment with cluster of differentiation 137 (CD137) agonist or immune checkpoint blockade therapies, anti-programmed-death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibody
* Severe infection within 4 weeks prior to randomization
* Significant history of cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Independent Review Facility (IRF)-Assessed Event Free Survival (EFS) | Up to approximately 96 months
  IRF-assessed EFS is defined as the time from randomization to the first documented disease progression per RECIST v1.1 that precludes surgery, local or distant disease recurrence, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | At time of surgery
  pCR is defined as the absence of any viable primary tumor cells at the time of surgical resection in the primary tumor and all sampled lymph nodes as assessed by central and local pathology laboratory.
Major Pathological Response (MPR) | At time of surgery
  MPR is defined as ≤ 10% residual viable tumor cells at the time of surgical resection in the primary tumor, as assessed by central and local pathology laboratory.
Objective Response (OR) | Prior to surgery, up to approximately 84 days
  Objective response is defined as a complete response or partial response, as determined by the investigator according to RECIST v1.1
Overall Survival (OS) | Up to approximately 96 months
  OS is defined as the time from randomization to death from any cause during the course of the study.
Investigator-Assessed EFS | Up to approximately 96 months
  EFS is defined as the time from randomization to the first documented disease progression per RECIST v1.1 that precludes surgery, local or distant disease recurrence, as assessed by the investigator; or death from any cause, whichever occurs first.
Disease-Free Survival (DFS) | Up to approximately 96 months
  DFS is defined as the time from the first date of no disease to local or distant recurrence (including occurrence of new primary NSCLC) or death due to any cause, whichever occurs first, as determined by the investigator during the adjuvant treatment and observation follow-up
2-Year and 3-Year OS | Up to approximately 96 months
  The 2-year and 3-year OS rate is defined as the probability that a participant will be alive 2 years and 3 years after randomization, respectively.
2-Year and 3-Year Independent Review Facility-Assessed EFS | Up to approximately 96 months
  EFS is defined as the probability that a participant will be event-free 2 years and 3 years after randomization, respectively, as assessed by the Independent Review Facility.
2-Year and 3-Year Investigator-Assessed EFS | Up to approximately 96 months
  EFS is defined as the probability that a participant will be event-free 2 years and 3 years after randomization, respectively, as assessed by the Investigator.
Change from baseline in HRQoL scores | Up to approximately 96 months
  Change from baseline in HRQoL scores as assessed through use of the two-item GHS/HRQoL subscale (Questions 29 and 30) of the EORTC QLQ-C30 at each assessment time point during the study through the completion of adjuvant treatment and observation follow-up assessments
Percentage of Participants With Adverse Events (AEs) | Up to approximately 96 months
Number and Severity of Surgical Related Adverse Events | Up to approximately 96 months
Number of Surgical Delays | Up to approximately 96 months
  Number of surgical delays.
Length of Surgical Delays | Up to approximately 96 months
  Length of surgical delays.
Number of Operative and Post-Operative Complications | Up to approximately 96 months
  Number of operative and post-operative complications.
Reasons for Surgical Cancellations | Up to approximately 96 months
  Reasons for surgical cancellations.
Minimum Observed Serum Atezolizumab Concentration (Cmin) | Pre-dose on Day 1 of Cycles 1 and 3 (each cylce is 21 days) for Neoadjuvant Treatment; pre-dose on Day 1 of Cycles 5, 7, 9, 11 and 19 (each cycle is 21 days) for Arm A; at treatment or observation follow-up discontinuation (up to approximately 96 months)
  Cmin is the minimum (or trough) concentration that a study drug achieves in the body.
Maximum Observed Serum Atezolizumab Concentration (Cmax) | Pre-dose on Day 1 of Cycles 1 and 3 for Neoadjuvant Treatment; Pre-dose on Day 1 of Cycles 5, 7, 9, 11 and 19 for Arm A. Each cycle is 21 days; at treatment or observation follow-up discontinuation (up to approximately 96 months)
  Cmax is the maximum (or peak) concentration that a study drug achieves in the body.
Percentage of Participants With Anti-Drug Antibody (ADA) to Atezolizumab | Pre-dose on Day 1 of Cycles 1 and 3 for Neoadjuvant Treatment; Pre-dose on Day 1 of Cycles 5, 7, 9, 11 and 19 for Arm A. Each cycle is 21 days; at treatment or observation follow-up discontinuation (up to approximately 96 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (122):
- United States (29):
  - Arizona Oncology, Tucson, Arizona
  - USC Norris Cancer Center, Los Angeles, California
  - The Center for Cancer Prevention and Treatment at St.Joseph Hospital of Orange, Orange, California
  - UC Davis Cancer Center, Sacramento, California
  - Scripps Clinic, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Illinois Cancer Care, Peoria, Illinois
  - Uni of Maryland Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Brighton Center for Specialty Care, Brighton, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Mercy Clinic Cancer & Hematology, Springfield, Missouri
  - Nebraska Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Northwell Health, Lake Success, New York
  - NYU Winthrop Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - South Austin, Austin, Texas
  - UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
- Australia (3):
  - St George Hospital, Kogarah, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Center, Melbourne, Victoria
- Austria (4):
  - Kepler Universitätskliniken GmbH - Med Campus III, Linz
  - Ordensklinikum Linz Elisabethinen, Linz
  - Klinik Penzing, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Brazil (3):
  - Cenantron - Centro Avancado de Tratamento Oncologico, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Shanghai Chest Hospital, Shanghai, China
- France (6):
  - CHU Angers, Angers
  - Centre Léon Bérard, Lyon
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Centre Hospitalier Saint Quentin, Saint-Quentin
  - CHU Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Hôpital d'Instruction des Armées de Sainte Anne, Toulon
- Germany (8):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios-Fachkliniken Muenchen-Gauting, Gauting
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Pius-Hospital Oldenburg, Oldenburg
  - Klinikum der Univer Regenburg, Regensburg
  - Robert Bosch Krankenhaus, Stuttgart
  - Missionsärztliche Klinik, Gemeinnützige Gesellschaft mbH, Würzburg
- Semmelweis Egyetem X, Budapest, Hungary
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Sourasky / Ichilov Hospital, Tel Aviv
- Italy (5):
  - Policlinico Universitario Campus Biomedico, Rome, Lazio
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - A.O. Universitaria Pisana-Ospedale Cisanello, Pisa, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- Japan (17):
  - Aichi Cancer Center Hospital, Aichi
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Kobe University Hospital, Hyōgo
  - Hyogo Medical University Hospital, Hyōgo
  - Kyoto University Hospital, Kyoto
  - Fukushima Medical University Hospital, Miyagi
  - Sendai Kousei Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - Kurashiki Central Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Krakowski Szpital Specjalistyczny im sw. Jana Paw?a II, Krakow
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad, Warsaw
- Russia (4):
  - Main Military Clinical Hospital named after N.N. Burdenko, Moscow, Moscow Oblast
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow, Moscow Oblast
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute named after N.N. Petrov, Saint Petersburg, Sankt-Peterburg
- University Hospital Medical Center Bezanijska kosa, Belgrade, Serbia
- University Clinic Golnik, Golnik, Slovenia
- South Africa (2):
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Eugene Marais Hospital, Pretoria
- South Korea (5):
  - Kosin University Gospel Hospital, Busan
  - St. Vincent's Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (10):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario la Fe, Valencia
- Sweden (4):
  - Lungmedicinska kliniken, Centrum för kirurgi, ortopedi och cancervård, Universitetssjukhuset, Linköping
  - Uni Hospital in Lund, Lund
  - Karolinska Universitetssjukhuset, Solna, Solna
  - Uppsala University Hospital, Uppsala
- Switzerland (2):
  - CHUV, Lausanne
  - UniversitätsSpital Zürich, Zurich
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Taichung Veterans General Hospital, Xitun Dist.
- Thailand (2):
  - Chulalongkorn Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk, Ukraine
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Barts and the London NHS Trust., London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Romero Roman A, Campo-Canaveral de la Cruz JL, Macia I, Escobar Campuzano I, Figueroa Almanzar S, Delgado Roel M, Galvez Munoz C, Garcia Fontan EM, Muguruza Trueba I, Romero Vielva L, Cano Garcia JR, Martinez Tellez E, Partida Gonzalez C, Jimenez Lopez MF, Jimenez Maestre U, Mongil Poce R, Sanchez Lorente D, Alvarez Kindelan A, Provencio Pulla M. Outcomes of surgical resection after neoadjuvant chemoimmunotherapy in locally advanced stage IIIA non-small-cell lung cancer. Eur J Cardiothorac Surg. 2021 Jul 14;60(1):81-88. doi: 10.1093/ejcts/ezab007. PMID 33661301